CLINICAL TRIAL: NCT03802968
Title: The Perioperative Application of Lung Ultrasound Combine With Diaphragm Ultrasound In One-lung Ventilation During Thoracic Surgery
Brief Title: The Application of Lung Ultrasound Combine With Diaphragm Ultrasound During Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-185
Record Dates: First submitted 2019-01-02; First posted 2019-01-14 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Videoassisted Thoracoscopic Surgery,One-lung Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perioperative lung-protective strategies had been advocated in one-lung ventilation but normal respiratory functions were yet impacted during videoassisted thoracoscopic(VATS) surgery. The primary aim of this study was to investigate respiratory complications after OLVby using bedside lung ultrasonography combine with diaphragmatic ultrasonography.

DETAILED DESCRIPTION:
Perioperative lung-protective strategies had been advocated in One-lung Ventilation(OLV) of videoassisted thoracoscopic(VATS) surgery but normal respiratory functions were yet impacted during general anesthesia, mechanical ventilation, loss of respiratory muscle tone and intrathoracic surgery. Lung ultrasonography has been confirmed to be a available tool for rapid confirming atelectasis, pleural effusion , pneumonia and pneumothorax. Diaphragmatic excursion were well correlated with vital capacity by lung function testing and diaphragmatic ultrasound imaging was demonstrated accurately to identify atrophy and impaired contractility or motion of the diaphragm.The primary aim of this present study was to investigate respiratory complications after OLV in the postoperative period by using bedside lung ultrasonography.The secondary aim was to evaluate the variation of lung ventilation during thoracoscopic surgery through lung ultrasonography combine with diaphragm ultrasound and assess the accuracy of ultrasound to confirm proper endobronchial intubation.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective thoracoscopic surgery of OLV, over 18 years of age

Exclusion Criteria:

* noncooperate from schizophrenia or delirium, a BMI higher than 40 kg/m2, a history of respiratory infection, a history of chronic obstructive pulmonary disease(COPD), a history of Chronic Heart Disease(CHD), received brachial plexus nerve block or general anesthesia within 2 weeks before surgery , received former thoracic procedures (e.g.,thoracotomy, thoracoscopy or thoracic drain)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective thoracoscopic surgery of OLV and over 18 years of age were included in the present study if they screened for the inclusion criteria. Patients were excluded if there were noncooperate from schizophrenia or delirium, a body mass index(BMI) higher than 40 kg/m2, a history of respiratory infection, chronic obstructive pulmonary disease(COPD), Chronic Heart Disease(CHD). Those received brachial plexus nerve block or general anesthesia within 2 weeks before surgery were also excluded. Former thoracic procedures (e.g.,thoracotomy, thoracoscopy or thoracic drain) were either criterions for exclusion.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Rate of respiratory complications after one-lung ventiltion(OLV) in the postoperative period by using bedside lung ultrasonography | 15 minutes after tracheal extubation

SECONDARY OUTCOMES:
The variation of lung ventilation during thoracoscopic surgery through lung ultrasound combined with diaphragm ultrasound | before induction, 5 minutes after intubation, 5 minutes after surgery,15 minutes after tracheal extubation

OTHER OUTCOMES:
Accuracy of Lung ultrasound in confirming proper endobronchial intubation | 5 minutes after one- lung ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Chair — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No